CLINICAL TRIAL: NCT03097965
Title: Safety Evaluation of a Lifestyle Modification Program for Healthy Weight and Cardiometabolic Function
Brief Title: Safety Evaluation of a Lifestyle Modification Program In.Form 1.1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nature's Sunshine Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSP-CT-004
Record Dates: First submitted 2017-03-14; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIET (Active Comparator): * High Phyto-PRO food plan
  * Physical activity
  * Cognitive behavioral program
  Interventions: Other: DIET
- PROGRAM (Experimental): * High Phyto-PRO food plan
  * Physical activity
  * Cognitive Behavioral Program
  * Protein Shakes
  * Phytosterols supplement
  * Berberine supplement
  * Anti-oxidant supplement
  * Probiotic supplement
  * Fish Oil supplement
  * Multiple Vitamin/Multiple Mineral supplement
  Interventions: Dietary Supplement: PROGRAM; Other: DIET

INTERVENTIONS:
Dietary Supplement: PROGRAM
  Arms: PROGRAM
Other: DIET

SUMMARY:
The study evaluated and compared the safety, tolerance and acceptability of a lifestyle modification program with or without nutritional supplementation in generally healthy overweight subjects with cardiometabolic risk factors.

DETAILED DESCRIPTION:
To investigate the safety, tolerance and acceptability of a low-glycemic load diet combined with exercise and lifestyle modification education (DIET) or a similar program with a meal replacement formula and targeted nutraceuticals (PROG) in generally healthy, overweight subjects, forty to fifty subjects with two or more cardiometabolic risk factors, aged 18 to 69 will be randomized into different arms, 13-week intervention trial. To evaluate safety and tolerability, questionnaires were collected weekly. Additionally, baseline, week 9 and 13 fasting blood samples will be drawn for blood counts, metabolic profiles, plasma lipids, and additional cardiovascular risk factors. Vitals signs, weight and body composition were monitored weekly.

ELIGIBILITY:
Inclusion Criteria:

Generally healthy subjects (men and women ≥ 18 and ≤ 69 years old) were required:

* to be overweight or obese (BMI ≥ 27 kg/m2 and ≤ 50 kg/m2),
* to exhibit visceral obesity (waist circumference ≥ 35 inches for women and ≥ 39 inches for men),
* and demonstrate signs of cardiometabolic dysfunction. Specifically, subjects were required to have:
* elevated LDL cholesterol ≥ 130 mg/dl
* and/or elevated TG defined as TG ≥ 130 mg/dl. Additionally, subjects were required to have at least one of the following criteria (unless subject had both elevated LDL and TG):
* HDL < 50 mg/dl for women and < 40 mg/dl for men,
* blood glucose ≥ 100 mg/dl, HbA1C ≥ 5.7%,
* or Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) score defined as ≥ 2.0.

Exclusion Criteria included:

* Pregnancy
* Lactation
* Recent changes in prescription medications, over-the-counter medications, medical foods, and nutritional supplements
* Recent or regular use of narcotics, investigational drugs, corticosteroids, anticoagulants, neuroactive medications, or medication or supplements relevant to hyperglycemia or hyperlipidemia
* Chronic use of over-the-counter medication which would interfere with study endpoints including NSAIDS, laxatives and antacids
* Allergy or intolerance to study products
* Serious, unstable medical conditions including known infection with HIV, tuberculosis or hepatitis; cardiovascular disease; Diabetes Mellitus; autoimmune diseases; malignancy; psychiatric disease; substance abuse;
* Abnormal laboratory findings
* Participating in or planning to begin a weight loss diet during the study period
* Difficulty in swallowing pills
* Lifestyle or schedule incompatible with the study protocol.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0". | 13 weeks
  Data collection including questionnaires at individual and group visits and physician interviews at individual visits (baseline, week 9 and week 13) will be used to assess participants for treatment-related adverse events.

SECONDARY OUTCOMES:
Number of participants with treatment-related changes in basic safety labs | 13 weeks
  Phlebotomy will be conducted at individual visits (baseline, week 9 and week 13). Comprehensive Metabolic Panels and Complete Blood Counts will be assessed for treatment-related change from baseline.
Number of participants with treatment-related changes in vital signs | 13 weeks
  Blood pressure and peripheral pulse will be monitored at individual visits (baseline, week 9 and week 13). Collected data will be assessed for treatment-related change from baseline.
Change in weight in pounds compared to baseline | 13 weeks
  Weight in pounds will be monitored (Tanita body composition monitor) at individual visits (baseline, week 9 and week 13) and group visits. Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in body fat in percentage compared to baseline | 13 weeks
  Body fat in percentage will be monitored (Tanita body composition monitor) at individual visits (baseline, week 9 and week 13) and group visits. Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in BMI in kg/m2 compared to baseline | 13 weeks
  BMI in kg/m2 will be monitored (Tanita body composition monitor) at individual visits (baseline, week 9 and week 13) and group visits. Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in waist circumference in inches compared to baseline | 13 weeks
  Waist circumference in inches will be monitored at individual visits (baseline, week 9 and week 13). Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in Total Cholesterol in mg/dl compared to baseline | 13 weeks
  Total Cholesterol in mg/dl will be measured at individual visits (baseline, week 9 and week 13). Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in LDL-Cholesterol in mg/dl compared to baseline | 13 weeks
  LDL-Cholesterol in mg/dl will be measured at individual visits (baseline, week 9 and week 13). Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in oxidized LDL-Cholesterol in mg/dl compared to baseline | 13 weeks
  Oxidized LDL-Cholesterol in mg/dl will be measured at individual visits (baseline, week 9 and week 13). Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in HDL-Cholesterol in mg/dl compared to baseline | 13 weeks
  HDL-Cholesterol in mg/dl will be measured at individual visits (baseline, week 9 and week 13). Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in fasting glucose in mg/dl compared to baseline | 13 weeks
  Fasting glucose in mg/dl will be measured at individual visits (baseline, week 9 and week 13). Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in fasting insulin in mIU/l compared to baseline | 13 weeks
  Fasting insulin in mIU/l will be measured at individual visits (baseline, week 9 and week 13). Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in Hemoglobin A1c in percentage compared to baseline | 13 weeks
  Hemoglobin A1c in percentage will be measured at individual visits (baseline, week 9 and week 13). Collected data will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in Metabolic Syndrome Score compared to baseline | 13 weeks
  A Metabolic Syndrome score (0-5) will be calculated for participants at individual visits (baseline, week 9 and week 13). The five features of Metabolic Syndrome (visceral adiposity based on waist circumference, hyperglycemia, hypertension (or use of antihypertensives), hypertriglyceridemia and low HDL-Cholesterol will each be assigned a point value of 1. Subjects will receive 1 point for each feature they demonstrate on collected data. Score will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.
Change in Framingham Risk Assessment Score compared to baseline | 13 weeks
  The Framingham Risk Assessment Score will be calculated for participants at individual visits (baseline, week 9 and week 13). Score will be assessed for treatment-related change from baseline. Comparison will be made between DIET and PROGRAM arms.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Lamb, MD, Principal Investigator — Hughes Center for Research and Innovation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahlberg CJ, Ou JJ, Babish JG, Lamb JJ, Eliason S, Brabazon H, Gao W, Kaadige MR, Tripp ML. A 13-week low glycemic load diet and lifestyle modification program combining low glycemic load protein shakes and targeted nutraceuticals improved weight loss and cardio-metabolic risk factors. Can J Physiol Pharmacol. 2017 Dec;95(12):1414-1425. doi: 10.1139/cjpp-2016-0704. Epub 2017 Aug 11. PMID 28800398